CLINICAL TRIAL: NCT06191913
Title: Assessment of Microcirculatory Alteration by a Vascular Occlusion Test Using Near-infrared Spectroscopy in Pediatric Cardiac Surgery:Effect of Cardiopulmonary Bypass
Brief Title: Microcirculatory Alteration by a Vascular Occlusion Test Using Near-infrared Spectroscopy in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, mustafa emre gürcü, Anesthesiology and reanimation, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2020/10/364
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Microcirculation
Keywords: Microcirculation; Vascular occlusion test; Near-infrared spectroscopy; Pediatric cardiopulmonary bypass; Congenital cardiac surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Near-infrared spectroscop — Before the induction of anesthesia, INVOS pediatric SomaSensor probe (Coviden, Dublin, Ireland) was placed on the patient's forearm and then connected to a monitor, which was used to continuously measure and assess the dynamic changes in the StO2
  Other Names: INVOS pediatric SomaSensor probe (Coviden, Dublin, Ireland)

SUMMARY:
Cardiopulmonary bypass cause microcirculatory alterations. Near infrared spectroscopic measurement of tissue oxygen saturation and vascular occlusion test are novel technologies for assessing the microcirculatory function of peripheral tissue specifically in patients undergoing cardiac surgery with cardiopulmonary bypass

DETAILED DESCRIPTION:
Cardiac surgery and cardiopulmonary bypass (CPB) procedures cause microcirculatory alterations, and microvascular alterations and the impairment of tissue oxygen saturation (StO2) after cardiac surgery with CPB have been associated with adverse patient outcomes. It has been shown that contact with foreign surfaces causes transient microcirculatory dysfunction and activation of the inflammatory and hemostatic systems and that tissue trauma and anesthesia also affect microcirculation. Although microcirculation is affected by surgery with CPB, monitoring of the microcirculatory function is still not part of routine practice. Continuous real-time monitoring may aid in the early detection of tissue malperfusion.

StO2 measurement using NIRS and vascular occlusion testing (VOT) are novel techniques for assessing the microcirculatory function of peripheral tissue, specifically in patients undergoing cardiac surgery with CPB. The level of StO2 is determined by the amount of oxygen delivered and consumed. The deoxygenation rate, minimum rSO2, and reoxygenation rate measured using VOT may indicate tissue perfusion, the local metabolic rate, the oxygen reserve, and microvascular reactivity. It has been shown that prolonged exposure to CPB is associated with abnormal vasomotor responses and end-organ dysfunction. Although the INVOS system is not commonly used for VOT in children undergoing cardiac surgery with CPB, we hypothesized that using this noninvasive method to measure StO2 would allow detection of the local metabolic rate and local tissue perfusion adequacy change and that StO2 changes would reflect the preexisting cardiovascular reserve.

ELIGIBILITY:
Inclusion Criteria:

Elective cardiac surgery with CPB

Exclusion Criteria:

* Skin and peripheral vascular disease,
* Taking medicine for vascular disease,
* Emergency procedures

Ages: 3 Months to 3 Years | Sex: All
Age Groups: Child
Study Population: 120 pediatric patients scheduled for elective cardiac surgery with CPB were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Dynamic changes in the StO2 | during operation
  The following VOT parameters were calculated: baseline StO2 (%), occlusion slope (%/min) from baseline until nadir, minimum StO2 (%), reperfusion slope (%/min) from the minimum value to the maximum value, reperfusion time (min) from cuff release to the maximum value, and maximum StO2 (%). VOT was performed five times: before induction of anesthesia (T1), after induction of anesthesia (T2), during the CPB with full flow (T3), after the termination of the CPB (T4), and after sternum closure (T5

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Emre Gurcu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savluk OF, Yilmaz AA, Yavuz Y, Arisut S, Ukil Isildak F, Turkmen Karaagac A, Ozbek B, Cine N, Tuncer E, Ceyran H. Assessment of microcirculatory alteration by a vascular occlusion test using near-infrared spectroscopy in pediatric cardiac surgery: effect of cardiopulmonary bypass. Expert Rev Med Devices. 2024 Mar;21(3):249-255. doi: 10.1080/17434440.2024.2306155. Epub 2024 Jan 19. PMID 38217402